CLINICAL TRIAL: NCT06331182
Title: Comparison Between Role of Dexmedetomidine and Ketamine as an Adjuvant in External Oblique Intercostal Plane Block for Post Thoracotomy Pain: A Randomized Trial
Brief Title: Dexmedetomidine and Ketamine as an Adjuvant in External Oblique Intercostal Plane Block for Post Thoracotomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR552/2/24
Record Dates: First submitted 2024-03-17; First posted 2024-03-26 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Dexmedetomidine; Ketamine; External Oblique Intercostal Plane Block; Post Thoracotomy Pain
MeSH Terms: interventions — Ketamine; Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine group (Experimental): Patients will receive external oblique intercostal plane block using 29 ml bupivacaine 0.25% + 1 ml ketamine (50 mg) after induction of general anesthesia.
  Interventions: Drug: Ketamine; Drug: Bupivacaine
- Dex group (Experimental): Patients will receive external oblique intercostal plane block using 29 ml bupivacaine 0.25% + 1 ml dexmedetomidine 0.5 μg/kg after induction of general anesthesia.
  Interventions: Drug: Dexmedetomidine; Drug: Bupivacaine

INTERVENTIONS:
Drug: Ketamine — Patients will receive external oblique intercostal plane block using 29 ml bupivacaine 0.25% + 1 ml ketamine (50 mg) after induction of general anesthesia.
  Arms: Ketamine group
Drug: Dexmedetomidine — Patients will receive external oblique intercostal plane block using 29 ml bupivacaine 0.25% + 1 ml dexmedetomidine 0.5 μg/kg after induction of general anesthesia.
  Arms: Dex group
Drug: Bupivacaine — 29 ml bupivacaine 0.25%

SUMMARY:
The aim of this study is to compare the role of dexmedetomidine and ketamine as an adjuvant in external oblique intercostal plane block for post thoracotomy pain.

DETAILED DESCRIPTION:
Postsurgical pain in patients who have undergone open thoracotomy for lung cancer or other lung surgeries is known to be very severe.

As a result, this pain alters spontaneous breathing, delays postoperative recovery, and persists as chronic post-thoracotomy pain syndrome . Post-thoracotomy pain syndrome is relatively common and is seen in approximately 50% of patients after thoracotomy. It is a chronic condition, and about 30% of patients might still experience pain 4 to 5 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-III.
* Scheduled for open thoracotomy.

Exclusion Criteria:

* Patients with neurological or intellectual disability.
* Infection at the injection site.
* Opioid addiction.
* Allergic reaction to local anesthetics.
* Coagulation abnormalities.
* Drug abuse.
* Pregnancy.
* Severe liver and/or renal failure.
* Uncontrolled hypertension.
* Severe cardiovascular problems.
* Diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Time to the 1st rescue analgesia | 48 hours postoperative.
  A standardized analgesic regimen will be prescribed in the post-operative period. All patients will receive paracetamol 1 gm every 6 h as routine analgesia. Rescue analgesia of morphine will be given as 3 mg bolus if the numeric rating scale (NRS) > 3 to be repeated after 30 min if pain persists until the NRS < 4. NRS will be assessed at 0, 4, 8, 12, 18, 24, 36 and 48 h postoperatively.

SECONDARY OUTCOMES:
Intraoperative fentanyl consumption | Intraoperative
  Additional fentanyl bolus dosages of 1 µg/kg IV will be administered if heart rate or mean arterial blood pressure elevated more than 20% of the baseline (after exclusion of other causes than pain).
Total morphine consumption in the 1st 24hr and 48 hr | 48 hours postoperatively.
  Rescue analgesia of morphine will be given as 3 mg bolus if the numeric rating scale (NRS)> 3 to be repeated after 30 min if pain persists until the NRS < 4. NRS will be assessed at 0, 4, 8, 12, 18, 24, 36 and 48 h postoperatively.
  NRS (0 represents "no pain" while 10 represents "the worst pain imaginable")
Degree of pain | 48 hours postoperatively.
  Degree of pain will be assessed by the numeric rating scale (NRS). NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). It will be assessed at 0, 4, 8, 12, 18, 24, 36 and 48 h postoperatively.
Heart rate | Till the end of surgery.
  Heart rate will be recorded preoperative, before performing of block, and every 15 min till the end of surgery.
Mean arterial blood | Till the end of surgery.
  Mean arterial blood will be recorded preoperative, before performing of block, and every 15 min till the end of surgery.
The incidence of adverse events | 48 hours postoperative
  Adverse events such as pneumothorax, local anesthetic systemic toxicity (LAST), bradycardia, hypotension, nausea, vomiting, respiratory depression, or any other complication.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed S Elsharkawy, MD, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, ElGharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author

REFERENCES:
- [Derived] Moharam SA, ElSharkawy MS, Abdelhamid AS, Abdelbadie A, Kohaf NA, El Rahman Elgaria MA, Attia A, Elkashef AM. Dexmedetomidine versus ketamine as adjuvants in external oblique intercostal plane block for post thoracotomy pain: a randomised trial. BMC Anesthesiol. 2025 Nov 26;25(1):602. doi: 10.1186/s12871-025-03476-2. PMID 41299290